CLINICAL TRIAL: NCT05001009
Title: Improving Implementation of Outpatient Goals of Care Conversations for Veterans With Serious Illness
Brief Title: Goals of Care Conversations Study
Acronym: LSTDI
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Health Services Research
Other Study IDs: IIR 19-018; HX002935 (Other: eRA Project Ref)
Record Dates: First submitted 2021-08-02; First posted 2021-08-11 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Seriously Ill Patients; Cancer; Heart Failure; Interstitial Lung Disease; Chronic Obstructive Pulmonary Disease; End-stage Renal Disease; End-stage Liver Disease; Dementia
Keywords: implementation science; primary health care; advance care planning; patient care planning; palliative care; goals of care conversation; serious illness
MeSH Terms: conditions — Neoplasms; Heart Failure; Lung Diseases, Interstitial; Pulmonary Disease, Chronic Obstructive; Kidney Failure, Chronic; End Stage Liver Disease; Dementia

STUDY DESIGN:
Intervention Model Description: Sequential multiple-assignment randomized clinical trial (SMART)
Who Masked: Investigator
Masking Description: The primary outcome of goals of care conversation notes is determined by whether notes are entered into the electronic health record. The data manager queries the VA corporate data warehouse to determine if these notes are completed. Because the data manager can see who wrote the notes, the data manager is not blinded. However, the investigators do not expect the data manager to judge whether the notes were completed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- No then high patient engagement (Active Comparator): First stage: No patient engagement. Low intensity clinician training. Second stage (responders only): No patient engagement and high intensity clinician training.
  Second stage (non-responders only): High patient engagement and high intensity clinician training.
  Interventions: Behavioral: Clinician Implementation Strategy Stage 1: low intensity clinician training; Behavioral: Clinician Implementation Strategy Stage 2: high intensity clinician training; Behavioral: High patient engagement
- No then low patient engagement (Active Comparator): First stage: No patient engagement. Low intensity clinician training. Second stage (responders only): No patient engagement and high intensity clinician training.
  Second stage (non-responders only): Low intensity patient engagement and high intensity clinician training.
  Interventions: Behavioral: Clinician Implementation Strategy Stage 1: low intensity clinician training; Behavioral: Clinician Implementation Strategy Stage 2: high intensity clinician training; Behavioral: Low patient engagement
- Low then high patient engagement (Active Comparator): First stage: Low intensity patient engagement. Low intensity clinician training.
  Second stage (responders only): No patient engagement and high intensity clinician training.
  Second stage (non-responders only): High patient engagement and high intensity clinician training.
  Interventions: Behavioral: Clinician Implementation Strategy Stage 1: low intensity clinician training; Behavioral: Clinician Implementation Strategy Stage 2: high intensity clinician training; Behavioral: Low patient engagement; Behavioral: High patient engagement
- Low then low patient engagement (Active Comparator): First stage: Low patient engagement. Low intensity clinician training. Second stage (responders only): No patient engagement and high intensity clinician training.
  Second stage (non-responders only): Low intensity patient engagement and high intensity clinician training.
  Interventions: Behavioral: Clinician Implementation Strategy Stage 1: low intensity clinician training; Behavioral: Clinician Implementation Strategy Stage 2: high intensity clinician training; Behavioral: Low patient engagement

INTERVENTIONS:
Behavioral: Clinician Implementation Strategy Stage 1: low intensity clinician training — A "booster" of the established LSTDI implementation strategy. Clinicians will be presented with summary written/electronic materials on the LSTDI developed for the study. Online training options and when and how to complete goals of care conversations and documentation will be highlighted.
Behavioral: Clinician Implementation Strategy Stage 2: high intensity clinician training — This includes two components:
  1. Team facilitation to help the primary care team (advance practice provider, nurse, social worker) work together to create roles and responsibilities for accomplishing goals of care conversations with patients
  2. A patient list "trigger" of patients potentially eligible for goals of care conversations (the patient study population) will be sent to the primary care clinicians.
Behavioral: Low patient engagement — Patients will be sent information about goals of care conversations, including the PREPARE website.
  Other Names: PREPARE information and website
  Arms: Low then high patient engagement; Low then low patient engagement; No then low patient engagement
Behavioral: High patient engagement — Patients will be sent information about goals of care conversations, including the PREPARE website. Follow-up phone calls to discuss goals of care conversations and the PREPARE website will be made.
  Other Names: PREPARE information and website and phone call
  Arms: Low then high patient engagement; No then high patient engagement

SUMMARY:
The long term goal is to improve quality of care in Veterans with serious illnesses by aligning medical care with Veterans' goals and values. The objective of this study is to use a sequentially randomized trial to determine what implementation strategies are effective to increase early, outpatient goals of care conversations. The study will use interviews with and surveys of medical providers, patients, and caregivers, along with medical record data. This work is significant because it tests ways Veterans can express their goals and preferences for life sustaining treatments and have them honored.

DETAILED DESCRIPTION:
The aims of this study are as follows:

Aim 1. Use a clinician-level SMART in three VA health systems to determine the effectiveness of clinician and patient implementation strategies to improve the occurrence of documented goals of care conversations in Veterans with serious medical illness. Hypothesis 1 (first stage of the SMART): Compared to a low intensity clinician strategy alone, a low intensity clinician and patient strategy will lead to increased documentation of goals of care conversations. Hypothesis 2. Among those who do not respond to low intensity strategies, compared to a high intensity clinician strategy paired with a low intensity patient strategy, a high intensity clinician and patient strategy will lead to increased documentation of goals of care conversations.

Aim 2a. Identify the sequence of implementation strategies that leads to the overall greatest increase in documentation of goals of care conversations. Aim 2b (exploratory). Identify patient and clinician characteristics that modify the effect of sequences of implementation strategies on documentation of goals of care conversations.

Aim 3. Understand clinician and patient implementation strategy success or failure using a mixed method evaluation involving clinicians, leaders, patients, and caregivers.

ELIGIBILITY:
Inclusion Criteria:

CLINICIANS VA primary care advance practice clinicians (MDs, APRNs, PAs) at one of the three study sites able to complete goals of care conversation notes and orders. Advance practice clinicians will be eligible for randomization if they have at least 15 eligible patients without goals of care conversation notes at the start of stage 1 (to allow participating clinicians ample opportunities to write notes) and have written fewer than 4 goals of care conversation notes in the previous 6 months (to select clinicians who need improvement), and can potentially receive the planned implementation strategies, i.e., clinicians who regularly attend the Patient Aligned Care Team (PACT) team meetings.

PATIENTS

* Veteran enrolled in VHA health care in one of the three study sites who is a current patient of one of the eligible primary care clinicians
* Diagnosis of cancer, heart failure, interstitial lung disease, chronic obstructive pulmonary disease, end-stage renal disease, end-stage liver disease, and dementia
* Care Assessment Need score of > or equal to 90 using the one-year combined hospitalization/mortality variable

Exclusion Criteria:

PATIENTS

* Prisoner
* Pregnant
* under 18 years of age.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2022-09-13 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Percent of patients with a goals of care conversation note documented in Stage 2 | From the start of stage 2 to 9 months later
  Amongst patients attributed to a clinician who was randomized in Stage 2, whether or not a goals of care conversation note was written during Stage 2.

SECONDARY OUTCOMES:
Percent of patients with a goals of care conversation note documented in Stage 1 or 2 | From the start of stage 1 to 9 months after the start of stage 2
  Amongst all patients in the study, whether or not a goals of care conversation note was written during the study.
Percent of patients with a goals of care conversation note documented in Stage 1 | From the start of stage 1 to the beginning of stage 2 (approximately 8 months)
  Amongst all patients in the study, whether or not a goals of care conversation note was written during stage 1

CONTACTS AND LOCATIONS:
Overall Officials: David Bekelman, MD MPH, Principal Investigator — Rocky Mountain Regional VA Medical Center, Aurora, CO; Anne M Walling, MD PhD, Principal Investigator — VA Greater Los Angeles Healthcare System, West Los Angeles, CA
Locations (3):
- United States (3):
  - VA Palo Alto Health Care System, Palo Alto, CA, Palo Alto, California
  - VA Greater Los Angeles Healthcare System, West Los Angeles, CA, West Los Angeles, California
  - Rocky Mountain Regional VA Medical Center, Aurora, CO, Aurora, Colorado

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ha DM, Deng LR, Lange AV, Swigris JJ, Bekelman DB. Reliability, Validity, and Responsiveness of the DEG, a Three-Item Dyspnea Measure. J Gen Intern Med. 2022 Aug;37(10):2541-2547. doi: 10.1007/s11606-021-07307-1. Epub 2022 Jan 3. PMID 34981344
- [Background] Haverfield MC, Ma J, Walling A, Bekelman DB, Brown-Johnson C, Lo N, Lorenz KA, Giannitrapani KF. Communication processes in an advance care planning initiative: A socio-ecological perspective for service evaluation. Palliat Med. 2024 Dec;38(10):1134-1143. doi: 10.1177/02692163241277394. Epub 2024 Sep 10. PMID 39254148
- [Result] Bekelman DB, Giannitrapani K, Linn KA, Langner P, Sudore RL, Rabin B, Lorenz KA, Foglia M, Glickman A, Pawlikowski S, Sloan M, Gamboa RC, McCaa MD, Hines A, Walling AM. Increasing goals of care conversations in primary care: Study protocol for a cluster randomized, pragmatic, sequential multiple assignment randomized trial. Contemp Clin Trials. 2024 Oct;145:107643. doi: 10.1016/j.cct.2024.107643. Epub 2024 Jul 27. PMID 39074531